CLINICAL TRIAL: NCT04310007
Title: A Randomized Phase II Trial of Cabozantinib and Cabozantinib Plus Nivolumab Versus Standard Chemotherapy in Patients With Previously Treated Non-Squamous NSCLC
Brief Title: Testing the Addition of the Pill Chemotherapy, Cabozantinib, to the Standard Immune Therapy Nivolumab Compared to Standard Chemotherapy for Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01541; NCI-2020-01541 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5191 (Other: ECOG-ACRIN Cancer Research Group); EA5191 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Lung Non-Squamous Non-Small Cell Carcinoma; Recurrent Lung Non-Squamous Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling; cabozantinib; Docetaxel; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Nivolumab; Paclitaxel; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Step 1, Arm A (cabozantinib S-malate) (Experimental): Patients in Step 1, Arm A receive cabozantinib S-malate PO QD. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may continue to receive therapy after investigator-assessed RECIST 1.1 defined progression, including stable clinical and performance status and have potential for continued clinical benefit. Patients also undergo ECHO as clinically indicated, CT throughout the trial, and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test
- Step 1, Arm B (cabozantinib S-malate, nivolumab) (Experimental): Patients in Step 1, Arm B receive cabozantinib S-malate PO QD and nivolumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may continue to receive therapy after investigator-assessed RECIST 1.1 defined progression, including stable clinical and performance status and have potential for continued clinical benefit. Patients also undergo ECHO as clinically indicated, CT throughout the trial, and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Nivolumab
- Step 1, Arm C (standard chemotherapy) (Active Comparator): Patients in Step 1, Arm C receive ramucirumab IV over 30-60 minutes and docetaxel IV over 1 hour on day 1, or docetaxel IV over 1 hour on days 1 and 8, or gemcitabine hydrochloride IV on days 1 and 8, or paclitaxel IV over 3 hours on day 1, or nab-paclitaxel IV over 30 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity and at the discretion of the treating physician. Patients also undergo ECHO as clinically indicated, CT throughout the trial, and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Docetaxel; Procedure: Echocardiography Test; Drug: Gemcitabine Hydrochloride; Drug: Nab-paclitaxel; Drug: Paclitaxel; Biological: Ramucirumab
- Step 2, Arm Z (cabozantinib S-malate, nivolumab) (Experimental): Patients in Step 2, Arm Z receive cabozantinib S-malate PO QD and nivolumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may continue to receive therapy after investigator-assessed RECIST 1.1 defined progression, including stable clinical and performance status and have potential for continued clinical benefit. Patients also undergo ECHO as clinically indicated, CT throughout the trial, and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Step 1, Arm A (cabozantinib S-malate); Step 1, Arm B (cabozantinib S-malate, nivolumab); Step 2, Arm Z (cabozantinib S-malate, nivolumab)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP 56976; RP-56976; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Step 1, Arm C (standard chemotherapy)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Gemcitabine Hydrochloride — Given PO
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
  Arms: Step 1, Arm C (standard chemotherapy)
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
  Arms: Step 1, Arm C (standard chemotherapy)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Step 1, Arm B (cabozantinib S-malate, nivolumab); Step 2, Arm Z (cabozantinib S-malate, nivolumab)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Step 1, Arm C (standard chemotherapy)
Biological: Ramucirumab — Given IV
  Other Names: Anti-VEGFR-2 Fully Human Monoclonal Antibody IMC-1121B; Cyramza; IMC 1121B; IMC-1121B; IMC1121B; LY 3009806; LY-3009806; LY3009806; Monoclonal Antibody HGS-ETR2
  Arms: Step 1, Arm C (standard chemotherapy)

SUMMARY:
This phase II trial compares cabozantinib alone and the combination of cabozantinib and nivolumab to standard chemotherapy in the treatment of patients with non-squamous non-small cell lung cancer (NSCLC). Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ramucirumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as docetaxel, gemcitabine hydrochloride, paclitaxel, and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cabozantinib alone or in combination with nivolumab may be more effective than standard chemotherapy in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether cabozantinib alone, or the combination of nivolumab and cabozantinib, as compared to standard chemotherapy alone, extends progression-free survival (PFS) for this patient population with non squamous NSCLC.

SECONDARY OBJECTIVES:

I. To determine the overall survival for each arm of the trial. II. To evaluate the best overall radiographic response rate for each arm of the trial.

III. To evaluate and describe the toxicity profile of monotherapy with cabozantinib, and the combination of nivolumab and cabozantinib in this patient population with non-squamous NSCLC.

EXPLORATORY IMAGING OBJECTIVES:

I. To describe time point tumor response assessment, overall best response, progression-free survival and overall survival using the conventional Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria and the exploratory revised CHOI criteria with all measurements performed by the central review.

II. To compare the progression-free survival using the RECIST1.1 imaging response assessment measurements by site study personnel to those performed by central review.

EXPLORATORY CORRELATIVE OBJECTIVE:

I. To perform correlative biomarker research on tissue and blood biospecimens collected within this trial.

OUTLINE:

STEP 1: Patients are randomized to 1 of 3 arms.

ARM A: Patients receive cabozantinib S-malate orally (PO) once daily (QD). Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may continue to receive therapy after investigator-assessed RECIST 1.1 defined progression, including stable clinical and performance status and have potential for continued clinical benefit.

ARM B: Patients receive cabozantinib S-malate PO QD and nivolumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may continue to receive therapy after investigator-assessed RECIST 1.1 defined progression, including stable clinical and performance status and have potential for continued clinical benefit.

ARM C: Patients receive ramucirumab IV over 30-60 minutes and docetaxel IV over 1 hour on day 1, or docetaxel IV over 1 hour on days 1 and 8, or gemcitabine hydrochloride IV on days 1 and 8, or paclitaxel IV over 3 hours on day 1, or nab-paclitaxel IV over 30 minutes on days 1 and 8. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity and at the discretion of the treating physician.

STEP 2: Patients in Arm C experiencing disease progression are assigned to Arm Z.

ARM Z: Patients receive cabozantinib S-malate PO QD and nivolumab IV over 30 minutes on day 1. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may continue to receive therapy after investigator-assessed RECIST 1.1 defined progression, including stable clinical and performance status and have potential for continued clinical benefit.

Patients in all arms undergo echocardiogram (ECHO) as clinically indicated, computed tomography (CT) throughout the trial, and collection of blood on study.

After the completion of study treatment, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* RANDOMIZATION (STEP 1): Patient must be >= 18 years of age
* RANDOMIZATION (STEP 1): Patient must have pathologically confirmed non-squamous non-small cell lung carcinoma (NSCLC). Patients with NSCLC not otherwise specified (NOS) are eligible. Mixed tumors will be categorized by predominant cell type. If small cell elements are present, the patient is ineligible
* RANDOMIZATION (STEP 1): Patient must have metastatic stage IVA or IVB disease (includes M1a, M1b, and M1c), according to the 8th edition of the lung cancer TNM classification system. Recurrent metastatic NSCLC ineligible for curative therapy (in the treating investigator's opinion) is also allowed
* RANDOMIZATION (STEP 1): Patient's tumor must be known negative for EGFR tyrosine kinase inhibitor (TKI) sensitizing mutations (for example at a minimum, negative for EGFR Exon 19 deletions, EGFR exon 20 insertions, and Exon 21 L858R, L861Q mutations ) AND negative for ALK gene rearrangements (by fluorescence in situ hybridization [FISH], next generation sequencing [NGS], or immunohistochemistry [IHC]) by routine Clinical Laboratory Improvement Amendments (CLIA)- or Food and Drug Administration (FDA)-certified clinical testing methods. CLIA or FDA approved circulating tumor deoxyribonucleic acid (DNA) testing is acceptable as an alternative to tissue testing
* RANDOMIZATION (STEP 1): Patient must have radiographic and/or clinical progression (per local investigator assessment) following one, but only one, line of platinum-based chemotherapy AND one, but only one, line of prior checkpoint inhibitor (anti-PD-1 or PD-L1) immunotherapy, either concurrently or sequentially in either order. A minimum of two doses of prior immunotherapy is required. Only one prior line of therapy is allowed if patients received chemotherapy and immunotherapy together (patients may not receive subsequent single agent chemotherapy), and greater than two prior lines of therapy are not allowed.

  * NOTE: Lines of therapy are defined by clinical or radiographic progression. For patients with recurrent metastatic NSCLC following treatment for stage 1-3 NSCLC, platinum-based chemotherapy received within 12 months of recurrence and/or immunotherapy received within 6 months of recurrence will meet the requirement for prior chemotherapy and/or immunotherapy but subsequent receipt of more immunotherapy and/or platinum-based chemotherapy is also allowed.
  * NOTE: Prior anti-VEGF antibody therapy (ie bevacizumab) is allowed. Prior ipilimumab, or investigational agents not excluded below, in combination with the required prior therapies above are allowed.
  * NOTE: Prior receipt of one or two lines of targeted therapy for ROS1, RET, MET, BRAF, ERBB2/HER2, or KRAS G12C positive NSCLC is allowed and will not count toward the line of therapy limit. However, progression is still required after chemotherapy and immunotherapy as above. Patients with ROS1, RET, MET positive NSCLC are strongly encouraged to get appropriate targeted therapy (such as crizotinib, entrectinib, lorlatinib, selpercatinib, pralsetinib, capmatinib, tepotinib, or another investigational, off-label, or approved agent directed against ROS1, RET, or MET positive NSCLC) prior to participation and will be stratified.
  * NOTE: No prior predominantly VEGFR directed TKI therapy (such as cabozantinib, lenvatinib, or sitravantinib) is allowed, except for the agents named above.
* RANDOMIZATION (STEP 1): The investigator must document the intended chemotherapy regimen should their patient be randomized to Arm C (docetaxel and ramucirumab, OR single agent chemotherapy - docetaxel, gemcitabine, paclitaxel, nab-paclitaxel). The patient must not have received the selected chemotherapy agent previously for metastatic disease
* RANDOMIZATION (STEP 1): Any prior chemotherapy (based on administration schedule) must have been completed in greater than or equal to the following times prior to randomization:

  * FDA approved targeted oral therapy must be completed >= 1 week prior
  * Chemotherapy and/or immunotherapy must be completed >= 2 weeks prior
  * Prior investigational agents must be completed >= 4 weeks prior.
* RANDOMIZATION (STEP 1): Prior radiation therapy is allowed with a 2 week washout prior to randomization. Patient must not receive any systemic treatment with radionuclides within 6 weeks prior to randomization. Patient must have no clinically relevant ongoing complication from prior radiation therapy
* RANDOMIZATION (STEP 1): Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen (in the opinion of the treating physician) are eligible for this trial
* RANDOMIZATION (STEP 1): Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents (such as anthracycline or HER2-directed antibody therapy, but not prior checkpoint inhibitor therapy), must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients must be class 2B or better
* RANDOMIZATION (STEP 1): Patient must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must have met the eligibility criteria outlined above
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must have measurable disease as defined by RECIST v1.1. Measurements must be obtained within 4 weeks prior to randomization/registration
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must have recovered to equal to or less than grade 1 toxicities related to prior treatment, unless toxicities are clinically non significant and/or stable on supportive therapy (as determined by the treating physician)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Absolute neutrophil count >= 1,500/mcL (obtained within 2 weeks prior to randomization)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Platelets >= 100,000/mcL (obtained within 2 weeks prior to randomization)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Hemoglobin >= 9 g/dL (obtained within 2 weeks prior to randomization)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (for patients with Gilbert's disease total bilirubin must be =< 3 x ULN) (obtained within 2 weeks prior to randomization)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (obtained within 2 weeks prior to randomization)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Creatinine =< 1.5 x ULN OR calculated (Cockcroft-Gault formula) or measured creatinine clearance >= 50 mL/min/1.73m^2 (normalized to body surface area [BSA]) for patients with creatinine levels greater than 1.5 times the institutional normal creatinine =< 1.5 X ULN or creatinine clearance >= 50ml/min/1.73m^2 (obtained within 2 weeks prior to randomization)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not be pregnant or breast-feeding due to the unknown effects of cabozantinib and nivolumab on human development and for the potential risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization/registration to rule out pregnancy.
  * A patient of childbearing potential is anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 6 months after completion of treatment on the study
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have clinically significant gastrointestinal bleeding within 6 months prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have pulmonary hemorrhage or hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have active drug induced pneumonitis within 3 months prior to randomization. Prior immune mediated pneumonitis of grade 3 or 4 are not eligible regardless of time window
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have current radiographic evidence of tumor invading major blood vessel, evidence of tumor cavitation > 1 cm, evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or evidence of endotracheal or mainstem endobronchial tumor
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have peptic ulcer disease, known malabsorption syndrome, bowel obstruction or gastric outlet obstruction within 3 months prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have grade 3 or greater infection, or infection requiring intravenous systemic treatment within 14 days prior to randomization. Patients must be off antibiotics at the time of randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have serious non-healing wound/ulcer/bone fracture within 28 days prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have history of organ transplant
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have concurrent symptomatic untreated hypothyroidism
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have history of major surgery within 3 months prior to randomization, minor surgery within 28 days prior to randomization, other minor procedures within 7 days prior to randomization, or clinically relevant ongoing complications from prior procedures
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 160 mm Hg systolic, or > 100 mm Hg diastolic despite optimal antihypertensive treatment
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have unstable angina pectoris, clinically-significant cardiac arrhythmias, stroke (including transient ischemic attack [TIA]), or myocardial infarction within 6 months prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients must not have a diagnosis of deep vein thrombosis/pulmonary embolism (DVT/PE) within 6 months of randomization unless stable, asymptomatic, and treated with low-molecular-weight heparin (LMWH) or a permitted oral anticoagulant for at least 7 days before randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must not be receiving anticoagulants (i.e., warfarin, aspirin, clopidogrel) except:

  * Prophylactic use of low-dose aspirin (100 mg po daily or less) and/or low dose molecular weight heparin (LMWH) is permitted.
  * Therapeutic doses of low dose molecular weight heparin (LMWH) or specified direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban are allowed in patients without untreated brain metastases who are on a stable dose 7 days prior to study randomization, and without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must not receive strong CYP3A4 inducers (e.g., dexamethasone (> 1 mg daily dosing), phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort) within 7 days prior to randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must have corrected QT interval calculated by the Fridericia formula (QTcF) =< 500 msec within 28 days prior to Step 1 randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must be able to swallow tablets
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must not be on continuous systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days prior to randomization, with the following exceptions:

  * Inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
  * Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
  * Physiologic replacement doses of systemic corticosteroids are permitted, if < 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients with brain metastases are eligible as follows:

  * Previously treated brain metastases must have been treated with radiation > 2 weeks prior to randomization or surgery > 3 months prior to randomization OR
  * Untreated (active) brain metastases are allowed if they are clinically asymptomatic, < 1 cm, non-hemorrhagic, the patient is not on systemic anticoagulation, and the investigator believes that central nervous system (CNS) specific treatment is unlikely to be required during the first 3 months of study treatment.
  * NOTE: Symptomatic leptomeningeal disease is NOT allowed
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must not have known active autoimmune disease or known history of autoimmune disease for which recurrence may affect vital organ function or require immune suppressive treatment including systemic corticosteroids (e.g., immune-related neurologic disease, multiple sclerosis, autoimmune neuropathy, Guillain-Barre syndrome, etc.).
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients with known history of human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients with known history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral at time of randomization (suppressive therapy is allowed, if indicated)
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load at time of randomization
* RANDOMIZATION (STEP 1 - ALL TREATMENT ARMS): Patient must not have had any prior allergic reaction or hypersensitivity to study drug components or related drugs (multitargeted small molecule tyrosine kinase inhibitors or checkpoint inhibitor monoclonal antibodies)
* STEP 2 (CROSSOVER ARM Z): Patient must have met all eligibility requirements for Step 1 at time of registration to Step 1 to be eligible for Step 2
* STEP 2 (CROSSOVER ARM Z): Patient must have radiographic progressive disease per RECIST criteria after >= 2 cycles of therapy on Arm C. The scan showing progression must be completed within 6 weeks prior to Step 2 registration
* STEP 2 (CROSSOVER ARM Z): Patient must not have intervening anticancer treatment or major surgical procedure(s) between Step 1 and Step 2, except palliative radiation which was completed >= 1 week prior to registration to Step 2
* STEP 2 (CROSSOVER ARM Z): Patient may not have central nervous system progression, but patients with stable CNS disease are allowed
* STEP 2 (CROSSOVER ARM Z): Patient must have an ECOG performance status 0-2
* STEP 2 (CROSSOVER ARM Z): Patient must have recovered to equal to or less than grade 1 toxicities related to prior treatment, unless the adverse event(s) are clinically non significant and/or stable on supportive therapy (as determined by the treating physician)
* STEP 2 (CROSSOVER ARM Z): Absolute neutrophil count >= 1,500/mcL (obtained within 2 weeks prior to registration to Step 2)
* STEP 2 (CROSSOVER ARM Z): Platelets >= 100,000/mcL (obtained within 2 weeks prior to registration to Step 2)
* STEP 2 (CROSSOVER ARM Z): Hemoglobin >= 9 g/dL (obtained within 2 weeks prior to registration to Step 2)
* STEP 2 (CROSSOVER ARM Z): Total bilirubin =< 1.5 x institutional ULN (for patients with Gilbert's disease total bilirubin must be =< 3 x ULN) (obtained within 2 weeks prior to registration to Step 2)
* STEP 2 (CROSSOVER ARM Z): AST(SGOT) and ALT(SGPT) =< 2.5 x ULN (obtained within 2 weeks prior to registration to Step 2)
* STEP 2 (CROSSOVER ARM Z): Creatinine =< 1.5 x ULN OR calculated (Cockcroft-Gault formula) or measured creatinine clearance >= 50 mL/min/1.73m^2 (normalized to BSA) for patients with creatinine levels greater than 1.5 times the institutional normal creatinine =< 1.5 X ULN or creatinine clearance >= 50ml/min/1.73m^2 (obtained within 2 weeks prior to registration to Step 2)
* STEP 2 (CROSSOVER ARM Z): Patient must have corrected QT interval calculated by the Fridericia formula (QTcF) =< 500 ms within 28 days prior to Step 2 registration
* STEP 2 (CROSSOVER ARM Z): Patient must not have any intercurrent illness or disease complication that the investigator believes would limit the ability to safely tolerate the combination of cabozantinib and nivolumab
* STEP 2 (CROSSOVER ARM Z): Patient must not be pregnant or breast-feeding due to the unknown effects of cabozantinib and nivolumab on human development and for the potential risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration to Step 2 to rule out pregnancy.
  * A patient of childbearing potential is anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* STEP 2 (CROSSOVER ARM Z): Patients must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for 6 months after completion of treatment on the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) for patient population with non-squamous no-small cell lung cancer (NSCLC) | After 58 events (From time of randomization to documented disease progression [site review of imaging] or death from any cause, whichever occurs first)
  The final analysis of PFS will be performed when the full information of PFS is reached (i.e., 58 events for each of the two primary comparisons). The two primary comparisons of PFS will each use a logrank test stratified on the randomization stratification factors with a one-sided type I error rate of 10%. Estimates of PFS including medians and confidence intervals, will be calculated using the Kaplan-Meier method. Cox proportional hazards models, stratified, on the same factors, will be used to estimate the treatment hazard ratios. At the final analyses, in the event that both primary PFS comparisons of the combination of nivolumab with cabozantinib and cabozantinib alone versus the standard chemotherapy are statistically significant, PFS will be compared between the two experimental arms (combination of nivolumab with cabozantinib versus [vs.] cabozantinib alone), using a stratified log rank test with a one-sided type I error rate of 10%.

SECONDARY OUTCOMES:
Overall survival (OS) for each arm | From time of randomization to documented disease progression (site review of imaging) or death from any cause, whichever occurs first, assessed up to 3 years
  The final analysis of OS will be performed when the full information of PFS is reached (i.e., 58 events for each of the two primary comparisons). OS will be tested in a hierarchical fashion if the primary comparison of PFS between treatment arms is statistically significant, using a log rank test stratified on the randomization stratification factors with a one-sided type I error rate of 10%. Estimates of OS, including medians and confidence intervals, will be calculated using the Kaplan-Meier method. Cox proportional hazards models, stratified, on the same factors, will be used to estimate the treatment hazard ratios. OS will be further tested in a hierarchical fashion if the comparison of PFS between the two experimental arms is statistically significant. Point estimates of all endpoints will be accompanied by the corresponding two-sided 80% confidence intervals. Subset analyses of PFS and OS by treatment arm will be estimated and compared within subsets.
Best objective response for each arm | Every 6 weeks for the first year on study, and then every 12 weeks after year one
  Will be evaluated via Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Response rates (complete response [CR] + partial response [PR]) and toxicity will be compared using Fisher's exact tests with a one-sided type I error rate of 10%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes. Modeling procedures will implement backward selection; variables significant at the 0.10 level in the univariate setting will be chosen for inclusion in an initial full model, and at each step the least significant variable will be removed from the model. Only those covariates with p < 0.05 will remain in any final models, unless there are factors identified by the study team as crucial to model interpretation. Point estimates of all endpoints will be accompanied by the corresponding two-sided 80% confidence intervals.
Toxicity profile of monotherapy with cabozantinib, and the combination of nivolumab and cabozantinib | Up to 3 years after completion of study treatment
  Will be determined using the Common Terminology Criteria for Adverse Events (CTCAE) criteria. Response rates (complete response [CR] + pathologic response [PR]) and toxicity will be compared using Fisher's exact tests with a one-sided type I error rate of 10%; multivariable logistic regression modeling will be used to adjust for the effect of any covariates that are associated with these categorical outcomes. Modeling procedures will implement backward selection; variables significant at the 0.10 level in the univariate setting will be chosen for inclusion in an initial full model, and at each step the least significant variable will be removed from the model. Only those covariates with p < 0.05 will remain in any final models, unless there are factors identified by the study team as crucial to model interpretation. Point estimates of all endpoints will be accompanied by the corresponding two-sided 80% confidence intervals.

OTHER OUTCOMES:
The RECIST1.1 response at each time point | Every 6 weeks for the first year on study, and then every 12 weeks after year one
  The measurement of each time point will be performed using the revised CHOI criteria will be only applied to arms A and B, which will include anti-angiogenic therapy. Both the RECIST1.1 and revised CHOI criteria will assess the overall best response as CR, partial PR, stable disease (SD), or progressive disease (PD). Their concordance will be assessed using the weighted Cohen's kappa coefficient (k) with quadratic weights. As a rule of thumb, the level of concordance between the two criteria will be considered poor (k <0), slight (k 0-0.20), fair (k 0.21-0.40), moderate (k 0.41-0.60), substantial (k 0.61-0.80), and almost perfect (k 0.81 - 1).
Agreement between central view and site review in terms of progression-free survival | After the completion of study treatment
  The progression status and the progression time will be assessed in agreement. The progression status is a binary measurement and the agreement will be assessed using the Cohen's kappa coefficient. For progression time, will assess the temporal agreement using the method developed by Zeng et al.
Correlative biomarker research | After the completion of study treatment
  Correlative biomarker research will be performed on tissue and blood specimens collected within this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Joel W Neal, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (614):
- United States (614):
  - Veterans Administration Medical Center - Birmingham, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Washington Hospital, Fremont, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Methodist Jennie Edmundson Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Freeman Physician Group of Pittsburg, Pittsburg, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Owensboro Health Mitchell Memorial Cancer Center, Owensboro, Kentucky
  - Mercy Health - Paducah Cancer Center, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Saint Agnes Hospital, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Henry Ford River District Hospital, East China Township, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Henry Ford Saint John Hospital - Academic, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Breast, Grosse Pointe Woods, Michigan
  - Henry Ford Saint John Hospital - Van Elslander, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Henry Ford Warren Hospital - Breast Macomb, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Henry Ford Rochester Hospital, Rochester Hills, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford Madison Heights Hospital - Breast, Warren, Michigan
  - Henry Ford Warren Hospital - GLCMS, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health - Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health - Ely Clinic, Ely, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health - Moose Lake Clinic, Moose Lake, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Oncology Associates PC, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Glens Falls Hospital, Glens Falls, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - ECU Health Oncology Kenansville, Kenansville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - ECU Health Oncology Richlands, Richlands, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Saint Luke's Hospital-Quakertown Campus, Quakertown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Self Regional Healthcare, Greenwood, South Carolina
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT04310007/ICF_000.pdf